CLINICAL TRIAL: NCT05983653
Title: Evaluation of Arthrocentesis With and Without Platelet Rich Plasma Injection in Patients With Disc Displacement With Reduction.
Brief Title: Evaluation of Arthrocentesis With and Without PRP Injection in Patients With Disc Displacement With Reduction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammad Ibraheem Mahmoud Alhoor, Principal Investigator ,master degree candidiate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: arthrocentesis and PRP on TMJ
Record Dates: First submitted 2023-07-13; First posted 2023-08-09 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: TMJ Disc Disorder
Keywords: anterior disc displacment with reduction
MeSH Terms: interventions — Arthrocentesis

STUDY DESIGN:
Intervention Model Description: After medical and dental history then clinical examination. A preoperative panoramic radiograph was taken as a primary survey to exclude the presence of any lesion at the area of interest and an MRI to evaluate disc position infiltration of plain anesthesia was administered to anesthetizing the auriculotemporal, posterior deep temporal, and masseter nerves. Scrubbing and draping of the patient was carried out by using betadine. Drawn canthotragal line. two needle insertion points are marked. The first will be at a distance of 10 mm from the tragus and 2 mm below the cantotragal line. The second point will be 20 mm in front of the tragus and 10 mm below this line. Two 19 gauge needles are inserted in these 2 points(upper joint space) Normal saline 200 ml is injected into the superior joint space. The second needle acts as an outflow portal
  * in the 1 st study group: The lavage will be 150 ml of normal saline
  * in the 2 nd study group: The lavage will be 150 ml of normal saline +PRP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 150 ml of normal saline lavage (Active Comparator): in the first arm, 150 ml of normal saline lavage alone without PRP
  Interventions: Procedure: arthrocentesis without PRP
- 150 ml arthrocentesis with PRP (Active Comparator): in the second arm, 150 ml of normal saline arthrocentesis with PRP
  Interventions: Procedure: arthrocentesis with PRP

INTERVENTIONS:
Procedure: arthrocentesis without PRP — 150 ml arthrocentesis without PRP
  Arms: 150 ml of normal saline lavage
Procedure: arthrocentesis with PRP — 150 ml arthrocentesis with PRP
  Arms: 150 ml arthrocentesis with PRP

SUMMARY:
This study is aiming To evaluate the treatment effect (anti-inflammatory and healing ) of PRP with arthrocentesis versus arthrocentesis alone on the management of anterior disc displacement with reduction

DETAILED DESCRIPTION:
The main aim is to determine whether arthrocentesis with and without PRP will affect the treatment outcome of arthrocentesis , in relation to pain , mouth opening, and disc position . PICO

(P): population : patient with TMD and have clinical signs of disc displacement (I): Intervention: arthrocentesis with normal saline (C): Comparison: two groups 150 ml of normal saline lavage and 150 ml arthrocentesis with PRP (O):Outcome :

Interventions: All patients involved in this study will be divided in to two different groups, one group will receive arthrocentesis with PRP and other group received arthrocentesis only

A through medical and dental history followed by clinical examination was carried out for all patients. Clinical measurements were taken to ensure patient adherence to our initial inclusion criteria prior to further investigations. A preoperative digital panoramic radiograph with 1:1 magnification was taken for each patient as a primary survey in order to exclude the presence of any lesion at the area of interest and MRI to evaluate disc position

Intra operative procedures for 2 groups:

This clinical report describes 2 different manipulations of arthrocentesis with or without PRP

• In two group: infiltration of plain anesthesia was administered using mepivacaine HCl (3%) to anaesthetizing the auriculotemporal nerve followed by subcutaneous at side of needle insertion. Injection to control pain . Scrubbing and draping of the patient was carried out in a standard fashion using betadine surgical scrub.

A straight line is drawn from the medial portion of the ear tragus to the lateral corner of the eye. In this line, two needle insertion points are marked. The first, more posterior point will be at a distance of 10 mm from the tragus and 2 mm below the canthus tragus line. This is the approximate area of the maximum concavity of the glenoid fossa. The distance is about 25mm from skin to the centre of the joint space .The second point will be 20 mm in front of tragus and 10 mm below this same line.

This marking indicates the site of the eminence of the TMJ. After the points of insertion for the two needles have been marked, local anaesthetic is injected at the planned entrance points. Two 19 gauge needles are inserted in the anterior and posterior recesses of the upper joint space . Through one needle, normal saline 200 ml is injected into the superior joint space. The second needle acts as an outflow portal, which allows lavage of the joint cavity

* in the control group:
* in the 1 st study group: The lavage will be 150 ml of normal saline
* in the 2 nd study group: The lavage will be 150 ml of normal saline +PRP

Follow up Patients will be evaluated at day of arthrocentesis and weekly there after for the first month and then after 6 month. clinical assessment will be achieved postoperatively to calculate and assessment of maximum mouth opening , pain and disc position.

Recruitment:

1. Patients' data will be enrolled in database of the Outpatient clinics of the Department of Oral & maxillofacial surgery, Faculty of Dentistry, Cairo University
2. If there is a potential eligibility, the patient will be examined thoroughly as described before.
3. Consecutive sampling is done through screening of patients. This will continue until the target population is achieved.
4. Identifying and recruiting potential subjects is achieved through patient database Assignment of interventions

Allocation:

1. Randomization:

   assistant supervisor will carry out the randomization process using a software www.rand.org with a ratio of 1:1.
2. Allocation concealment mechanism:

   All patients who give consent for participation and who fulfill the inclusion criteria will be randomized. Funded patient files in a dark sealed envelope will be the method for allocation concealment.
3. Implementation The supervisors are responsible of division the sealed envelopes into four groups and implementation for patients allocation. Enrolling and helping participants to interventions will by researcher

   Masking/blinding:

   Each patient will be given a code by the researcher and the observers will be blind to which group this case belong. Patients, evaluators and statistician will be blinded.

   Data collection, management, and analysis:

   Data collection methods Primary Outcome: The researcher and assistant supervisor. will calculate and assessment of mouth opening , pain and jaw movement for TWO groups.

   Plans to promote participant retention and complete follow- up:

   Participant Retention:

   A periodic regular follow up recalls will be planned .

   Participant Withdrawal:

   The patient is allowed to drop at any time from the study Participant withdrawal will be recorded and the patient will be excluded from the study. A percentage in the sample size is calculated to make up for any losses. The investigator also may withdraw participants from the study under strict certain conditions and only if the proposed therapy were considered harmful to the patient.

   Data management:

   Data forms and data entry

   All these procedures will be done by Supervisor :

   All data will be entered electronically. Patient files are to be stored in numerical order and stored in secure and accessible place. All data will be maintained in storage for 1 year after completion of the study.

   The electronic data and the scans of the patient will be backed up on a Drop box file for ensuring back up and ease of accessibility. Data Transmission and editing The assessor data entry will be transmitted from the assessors to database officer in the blind separate datasheets who in return record them in participant chart before sending them to the statistician. Security and Back-up of data All forms of the procedures related to study data will be kept in the project secure folder. Access to the study data will be restricted only to database officer. A complete back up of the primary database will be performed twice a month. Back-ups of periodic data analysis file will be kept.

   Statistical methods:

   Data will be coded and entered using the statistical package SPSS version 22. Data will be summarized using mean and standard deviation. Data will be explored for normality using kolmogorov smirnov test. Comparisons between two groups for normally distributed data will be done using analysis of variance (ANOVA), while for non-normally distributed numeric variable will be done by kruskal wallis test. Categorical data will be analyzed using chi square test. P value less than or equal to 0.05 will be considered statistically significant. All test will be two tailed.

   Data monitoring:

   Monitoring The main supervisor will be responsible for data monitoring to evaluate the outcome measures and any possible side effects that might affect the outcome.

   Audit Auditing of the study design will be done by the assistant supervisor

   Ethics and dissemination

   Research ethics approval This protocol and the template informed consent form will be reviewed by the Ethics Committee of Scientific Research - Faculty of Dentistry - Cairo University

   Protocol amendments Any modifications to the protocol which may impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, sample sizes, study procedures, or significant administrative aspects will require a formal amendment to the protocol. Such amendment will be agreed upon by the Council of oral and maxillofacial surgery department.

   Informed consent Researcher M.A will introduce and discuss the trial to patients who will be shown a video regarding the main aspects of the trial. Patients will then be able to have an informed discussion with the participating consultant. Researcher will obtain written consent from patients willing to participate in the trial. All consent forms will be translated into Arabic.

   Confidentiality All study-related information such as photos, panoramic x-ray, forms, charts will be stored in a password protected folder on the department database. The password will be available to the study team. But any personal information related to the patient's ID will be stored in and will acquire a coded ID with access only to the database officer.

   Declaration of interest The study is self-funded and there is no conflict of interest to declare.

   Access to data All the research team will have access to the data sets. All data sets will be password protected. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information and the participant will be only identified by patient number.

   Post-trial care All patients will have the primary research contact number in case there is any emergency. Follow up will continue until all patients are satisfied.

   Dissemination policy Study results will be published as partial fulfillment of the requirements for master's degree in Oral and maxillofacial surgery. Topics suggested for presentation or publication will be circulated to the authors

ELIGIBILITY:
Inclusion Criteria:

Healthy adult participants were chosen to participate in this study according to predefined inclusion criteria Wilkes stage II (chronic pain with good range of motion of anterior disk displacement with reduction and patients with painful joint noises occurring during mouth opening and/or closing including the clinical and MRI findings of anterior disc displacement with reduction that not respond to conservative therapies).Willingness and ability to commit follow-up

Exclusion Criteria:

Patients were excluded from the study if they had previous TMJ surgery, a medical history of any systematic disease, and patients participating in other studies.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
TMJ pain | first day , after 1 week , after 1 month, 3 month and after 6 months of procedure
  pain will be measured by Numerical rating scale from 0-10 (0 the lowest pain , 10 the greatest pain) ,will be measured before intervention , immediately after intervention and on follow up ( 1 week , 1 month , 3 month and 6 month after intervention )

SECONDARY OUTCOMES:
maximum mouth opening | first day , after 1 week , after 1 month, 3 month and after 6 months of procedure
  maximum mouth opening will be measured by ruler (millimeter) ,will be measured before inervention , immediately after intervention and on follow up ( 1 week , 1 month, 3 month and 6 month after intervention )
Disc position on TMJ | before procedure and after 6 months of procedure
  Disc position will by Magnetic resonance imaging (MRI) assessment if their anterior disc displacement with reduction , before intervention and after 6 month of intervention for any improvement with disc position

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine AA Nassar, Study Director — Cairo University
Locations (1):
- Faculty of dentistry Cairo Universty, Cairo, Manial, Egypt

REFERENCES:
- [Background] Abbadi W, Kara Beit Z, Al-Khanati NM. Arthrocentesis, Injectable Platelet-Rich Plasma and Combination of Both Protocols of Temporomandibular Joint Disorders Management: A Single-Blinded Randomized Clinical Trial. Cureus. 2022 Nov 11;14(11):e31396. doi: 10.7759/cureus.31396. eCollection 2022 Nov. PMID 36523721